CLINICAL TRIAL: NCT07094893
Title: A Biomarker Enrichment Trial of Anti-EGFR Agents in Patients With Advanced Colorectal Cancer (aCRC) With Wild-type RAS and Right Primary Tumour Location (Right-PTL).
Brief Title: Anti-EGFR Agents in Patients With Right-sided Advanced Colorectal Cancer With Wild-type RAS and AREG/EREG High Status
Acronym: ARIEL-ENGIC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARIEL-ENGIC
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: metastatic colorectal cancer; first-line; right primary tumour location; AREG; EREG; RAS wild-type; anti-EGFR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doublet or Triplet +/- Bevacizumab (Active Comparator): FOLFOX or CAPOX or FOLFIRI or FOLFOXIRI +/- bevacizumab.
  Treatment regimen and the dosage of each product in both arms will be at Investigators' discretion and in accordance with European guidelines (ESMO).
  Chemotherapy backbone is at investigators' choice as per clinical practice and guidelines according to the labels of each IMP. Choice of regimen will depend upon individual patient characteristics and choices, as judged by their oncologist. The choice of adding or not bevacizumab will be at investigators' evaluation according to its label and after evaluating any contraindication to its administration. The study treatment consists of the first 16 weeks of 1st line induction chemotherapy, followed by continuation of chemotherapy +/- bevacizumab, maintenance treatment or treatment break as per investigator and patient preference.
  Interventions: Drug: Bevacizumab; Drug: Irinotecan (CPT-11); Drug: Oxaliplatin; Drug: Leucovorin and 5-FU; Drug: Capecitabine
- Doublet + Cetuximab (Experimental): FOLFOX or FOLFIRI + Cetuximab.
  Treatment regimen and the dosage of each product in both arms will be at Investigators' discretion and in accordance with European guidelines (ESMO).
  Chemotherapy backbone is at investigators' choice as per clinical practice and guidelines according to the labels of each IMP. The study treatment consists of the first 16 weeks of 1st line induction chemotherapy, followed by continuation of chemotherapy + cetuximab, maintenance treatment or treatment break as per investigator and patient preference.
  Interventions: Drug: Cetuximab (EGFR inhibitor); Drug: Irinotecan (CPT-11); Drug: Oxaliplatin; Drug: Leucovorin and 5-FU

INTERVENTIONS:
Drug: Cetuximab (EGFR inhibitor) — Administration according to the labels of each IMP.
  Arms: Doublet + Cetuximab
Drug: Bevacizumab — Administration according to the labels of each IMP.
  Arms: Doublet or Triplet +/- Bevacizumab
Drug: Irinotecan (CPT-11) — Administration according to the labels of each IMP.
Drug: Oxaliplatin — Administration according to the labels of each IMP.
Drug: Leucovorin and 5-FU — Administration according to the labels of each IMP.
Drug: Capecitabine — Administration according to the labels of each IMP.
  Arms: Doublet or Triplet +/- Bevacizumab

SUMMARY:
The aim of this trial is to assess the feasibility of EREG/AREG assessment as a clinical diagnostic standard, used to guide clinical decision making in right-PTL, RAS-wt aCRC. Further to this, the aim is to determine whether EREG/AREG status identifies right-PTL participants who will benefit from the addition of anti-EGFR therapy to first-line chemotherapy.

DETAILED DESCRIPTION:
ARIEL-ENGIC is a multi-centre, phase IV, open label, randomised controlled biomarker enrichment trial with an internal pilot phase in which participants with wild-type RAS, right-PTL and EREG/AREG high aCRC will be randomized in a 1:1 ratio to receive chemotherapy (doublet) plus cetuximab versus chemotherapy (doublet or triplet) alone or with bevacizumab.

ARIEL-ENGIC is an international trial in which the UK (recruitment ongoing) and EU (Italy, Germany and Spain) are participating. ARIEL-ENGIC aims to randomize 280 participants at a global level. In Europe 60 centers will be involved and 120 participants (40 pts per Member State involved) will be randomized.

Given the biomarker prevalence, 660 participants will be registered to identify sufficient RAS-wt participants with high tumour EREG/AREG expression.

The ARIEL-ENGIC study has 2 phases, registration and randomization (the main trial). Participants meeting all of the inclusion criteria and none of the exclusion criteria for registration will be considered for trial eligibility and biomarker analysis. Tumour samples will be sent for centralized biomarker (EREG/AREG) assessment. Participants with high tumour EREG/AREG will be eligible for randomisation. Participants eligible for the randomisation phase will be allocated 1:1 to chemotherapy alone or with bevacizumab or chemotherapy plus anti-EGFR agent.

Stratification factors will be:

* Choice of first-line chemotherapy (irinotecan-based doublet; oxaliplatin-based doublet; FOLFOXIRI)
* Tumour location (transverse vs caecum vs ascending)
* Prior adjuvant or neoadjuvant chemotherapy (yes vs no)
* Primary tumour resected
* Country of registration

ELIGIBILITY:
Inclusion Criteria for Registration:

* Age ≥18 years
* Biopsy-confirmed adenocarcinoma of the colon with a right primary tumour location
* aCRC defined as either M1 or locally inoperable disease
* Tumour RAS status either wild-type (by local testing) or unknown
* Fit for combination chemotherapy plus anti-EGFR agent
* Sufficient tumour material for EREG/AREG analysis
* Written informed consent for registration

Exclusion Criteria for Registration

* Tumour RAS-mutation present
* Prior chemotherapy for aCRC
* Prior anti-EGFR agent therapy

Inclusion Criteria for Randomisation:

* Registered in ARIEL-ENGIC
* Local testing confirms tumour RAS-wt status
* ARIEL-ENGIC central testing confirms tumour EREG/AREG high
* Tumour measurable by RECIST v1.1 criteria on CT scan
* Participants have had CT scan within the timeframes stipulated (If there is a contrast reaction, then non-contrast CT with MRI is acceptable, assuming at least one of these modalities shows measurable disease at baseline for ETS evaluation and both modalities are repeated at the trial timepoints at week 8 and 16 and every 8 weeks until disease progression.)
* Pre-randomisation laboratory tests :
* Neutrophils ≥1.5 x109/l and platelet count ≥100 x109/l
* Serum bilirubin ≤ 1.25 x upper limit of normal (ULN), alkaline phosphatase

  * 5x ULN, and serum transaminase (either AST or ALT) ≤ 2.5 x ULN
* Estimated creatinine clearance ≥50ml/min (creatinine clearance estimated as per local practice)
* WHO performance status (PS) 0, 1 or 2
* Fit for combination chemotherapy plus anti-EGFR agent
* Life expectancy of at least 12 weeks
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit.
* Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception
* Written informed consent for randomization.

Exclusion Criteria for Randomisation:

* Participant has received more than one cycle of chemotherapy since registration
* Participants with history of hypersensitivity to any component of their proposed trial treatment regimen or any of their excipients
* Participants in receipt of live vaccine within four weeks prior to randomisation
* Participants with a history interstitial pneumonitis/idiopathic lung disease (ILD) or pulmonary fibrosis
* Participants with a history of keratitis, ulcerative keratitis or severe dry eye
* Participants with a history of severe skin reaction which in the clinicians' opinion could be exacerbated by EGFR Mab (cf Steven's Johnson Syndrome)
* Complete dihydropyrimidine dehydrogenase (DPYD) deficiency
* Untreated brain metastases or spinal cord compression or primary brain tumours
* History or evidence upon physical examination of CNS disease unless adequately treated
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration
* Clinically significant (e.g. active) cardiovascular disease for example cerebrovascular accidents, myocardial infarction, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years that are likely to have an impact upon survival or treatment delivery
* Known human immunodeficiency virus (HIV)
* Has documented presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to enrolment
* Has a positive hepatitis C virus (HCV) antibody test result at screening or within 3 months prior to enrolment. Note: Participants with a positive HCV antibody test result due to prior resolved disease can be randomised, only if a confirmatory HCV RNA test is obtained - Definite contraindications for the use of corticosteroids and antihistamines as premedication.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Woman pregnant or lactating or expecting to conceive children within the projected duration of the study through 6 months after the last dose of bevacizumab and/or fluorouracil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Early tumour shrinkage (ETS) | 8 weeks after treatment start
  To determine whether first-line chemotherapy (doublet) with cetuximab is more effective than chemotherapy (doublet or triplet) with or without bevacizumab in achieving early tumour shrinkage (ETS) after 8 weeks of treatment in randomised patients.
Overall survival (OS) | 50 months
  To assess whether the effectiveness of first-line chemotherapy (doublet) with cetuximab is more effective than chemotherapy (doublet or triplet) with or without bevacizumab in terms of overall survival (OS).

SECONDARY OUTCOMES:
Depth of response (DpR) | 24 months
  Depth of response (DpR) is defined as the maximum tumour shrinkage of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline, assessed at 16 weeks from start of treatment.
Objective Response Rate (ORR) | 24 months
  Objective Response Rate (ORR) is defined as the percentage of participants, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the study treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS) is defined as the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for participants who are alive, on study and progression free at the time of the analysis. Alive participants who have no tumor assessments after baseline will have time to event censored on the date of randomization.
Overall Toxicity Rate | 24 months
  Overall Toxicity Rate is defined as the percentage of participants, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the treatment.
Toxicity Rate | 24 months
  Toxicity Rate is defined as the percentage of participants, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3 - 4, according to National Cancer Institute Common Toxicity Criteria (version 5.0)3, during the treatment.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Questionnaires will be administered at baseline, 8 weeks, 16 weeks, 12- and 24-months post-randomisation.
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. Raw scores are standardized and converted into scale scores ranging from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Module for Colorectal cancer 29 (EORTC QLQ-CR29). | Questionnaires will be administered at baseline, 8 weeks, 16 weeks, 12- and 24- months post-randomisation.
  The EORTC QLQ-CR29 includes 29 items that evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others) that are associated with CRC and its treatments. There are separate items for patients with and without a stoma and separate items to evaluate the sexual function of men and women. Raw scores are standardized and converted into scale scores ranging from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life - Additional items to cover anti-EGFR (IL126) | Questionnaires will be administered at baseline, 8 weeks, 16 weeks, 12- and 24- months post-randomisation.
  The EORTC IL126 includes 20 items that evaluate additional items to cover anti-EGFR symptomatic toxicity. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life EQ-5D-3L (3-level version of EQ-5D by the EuroQol Group) | Questionnaires will be administered at baseline, 8 weeks, 16 weeks, 12- and 24- months post-randomisation.
  The EQ-5D-3L consists of: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Cremolini, MD, PhD, Study Chair — Department of Translational Research and New Technologies in Medicine and Surgery, University of Pisa

IPD SHARING:
Plan to Share IPD: No